CLINICAL TRIAL: NCT01852994
Title: Exercise Training and Testosterone Replacement in Heart Failure Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Testosterone
Record Dates: First submitted 2013-03-11; First posted 2013-05-14 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2013-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — testosterone undecanoate; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise training (Other): Aerobic and strength exercise training
  Interventions: Other: Exercise training
- Testosterone replacement (Other): Testosterone replacement will be done quarterly
  Interventions: Drug: Testosterone replacement
- Testosterone replacement+Exercise (Other): Both Testosterone replacement and Exercise will done
  Interventions: Drug: Testosterone replacement; Other: Exercise training

INTERVENTIONS:
Drug: Testosterone replacement — Application quarterly of Testosterone Undecylate
  Other Names: Testosterone Undecylate (Nebido)
  Arms: Testosterone replacement; Testosterone replacement+Exercise
Other: Exercise training — Aerobic and strength exercise training
  Arms: Exercise training; Testosterone replacement+Exercise

SUMMARY:
The purpose of this study is to determine if exercise training with or without testosterone replacement can improve cardiopathy in heart failure patients

DETAILED DESCRIPTION:
In this study, we are evaluating:

* hospital length of stay and readmission
* muscle sympathetic nerve activity
* functional capacity
* body composition

ELIGIBILITY:
Inclusion Criteria:

* heart failure
* hypogonadism
* left ventricular fraction ejection < 45%

Exclusion Criteria:

* chronic renal failure
* normal testosterone
* pace maker

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Microneurography | 4 months of exercise training/testosterone replacement
  Muscle sympathetic nerve activity (MSNA) is recorded directly from the peroneal nerve using the microneurography technique. Multiunit postganglionic muscle sympathetic nerve recordings is made using a tungsten microelectrode. All of the recordings of MSNA met previously established and described criteria. MSNA is quantified as burst frequency (bursts per minute).
Forearm blood flow | 4 months of exercise training/testosterone replacement
  Forearm blood flow is measured by venous occlusion plethysmography. The nondominant arm is elevated above heart level to ensure adequate venous drainage. A mercury-filled silastic tube attached to a low-pressure transducer is placed around the forearm and connected to a plethysmography. Forearm blood flow is determined on the basis of a minimum off four separate readings. Forearm vascular conductance is calculated by dividing forearm blood flow by mean arterial pressure times 100 and expressed in arbitrary units.

SECONDARY OUTCOMES:
Cardiopulmonary exercise | 4 months of exercise training/testosterone replacement
  The maximal cardiopulmonary test is carried out on a bike using a ramp protocol with workload increment every minute with energetic demand of about 1 metabolic equivalent(MET) per minute or 3.5 mL/Kg.min of oxygen uptake.
Body composition | 4 months of exercise training/testosterone replacement
  Body composition and bone mineral density is determined by dual energy x-ray absorptiometry using densitometry equipment (Hologic), at the following regions: lumbar spine, femoral neck, total femur and total body. Appendicular lean mass is calculated as the sum of arms and legs lean soft tissue masses, assuming that all non-fat and non-bone tissue is skeletal muscle. The total body fat is expressed in grams and as a percentage of body weight.
Muscle biopsy | 4 months of exercise training/testosterone replacement
  The muscle biopsy is obtained with a single entry into the muscle 5-10 minutes after administering the local anesthetic following an incision through the skin. A portion of the muscle (~10 mg) is processed to evaluate 1) muscle fiber type and 2) cross-sectional area

CONTACTS AND LOCATIONS:
Overall Officials: Maria Janieire N Alves, MD; PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto do Coração do Hospital da Clínicas da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil